CLINICAL TRIAL: NCT02393144
Title: Analysis of Contemporary Labor Patterns Measured Via Transperineal Ultrasonography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Collaborators: Middle East Technical University (Other)
Responsible Party: Principal Investigator, Erkan Kalafat, Research Assistant, Ankara University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 001
Record Dates: First submitted 2015-02-22; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Pregnancy; Obstetric Labor
Keywords: Labor analysis; Transperineal ultrasound imaging; Labor curve
MeSH Terms: interventions — Cardiotocography; Amniotomy; Analgesics; Analgesics, Opioid; Meperidine; Oxytocin; Labor, Induced; Cervical Ripening; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spontaneous labor arm (Other): Women with term pregnancies whose labor started spontaneously. Spontaneous labor is determined by either spontaneous rupture of membranes at term and/or powerful, regular uterine contractions that cause cervical change. Women will be admitted to labor ward after initial assessment via transperineal ultrasonography. Labor augmentation will be performed for women with inadequate uterine contractions, i.e. contractions measuring less than Montevideo units, irregular weak uterine contractions. Analgesia will be provided via administration of 50 mg intramuscular meperidine at 2 hour intervals as required. Amniotomy will be performed for women with adequate cervical dilatation and fetal head-descent. Transperineal ultrasonography will be performed at irregular intervals to assess cervical dilatation, angle of progression and fetal head position. After birth, birth time, birth weight, APGAR scores, degree of perineal trauma, episiotomy use will be recorded.
  Interventions: Device: Transperineal ultrasonography, General Electric Healthcare Voluson Ultrasound System; Device: Cardiotocography, Bionet FC1400 Fetal Monitor; Other: Amniotomy; Drug: Analgesics, Opioid, Meperidine; Drug: Labor augmentation, Oxytocin
- Induced labor arm (Other): Women with term pregnancies who are induced for birth before the onset of spontaneous labor. Labor will be induced with either oxytocin infusion for women with high Bishop score, or labor will be induced with dinoprostone pessary for women requiring cervical ripening, i.e. poor. Women will be admitted to labor ward after initial assessment via transperineal ultrasonography. Analgesia will be provided via administration of 50 mg intramuscular meperidine at 2 hour intervals as required. Amniotomy will be performed for women with adequate cervical dilatation and fetal head-descent. Transperineal ultrasonography will be performed at irregular intervals to assess cervical dilatation, angle of progression and fetal head position. After birth, birth time, birth weight, APGAR scores, degree of perineal trauma, episiotomy use will be recorded.
  Interventions: Device: Transperineal ultrasonography, General Electric Healthcare Voluson Ultrasound System; Device: Cardiotocography, Bionet FC1400 Fetal Monitor; Other: Amniotomy; Drug: Analgesics, Opioid, Meperidine; Drug: Labor induction, Oxytocin; Drug: Cervical ripening, labor induction, Dinoprostone

INTERVENTIONS:
Device: Transperineal ultrasonography, General Electric Healthcare Voluson Ultrasound System — Assessment of cervical dilatation, angle of progression and head position via transperineal ultrasonography
Device: Cardiotocography, Bionet FC1400 Fetal Monitor — Assessment of strength of uterine contractions (Montevideo units) and fetal heart rate (beat per minute) with electronic monitors.
Other: Amniotomy — Artificial rupture of membranes to assess meconium staining and induce labor speed.
Drug: Analgesics, Opioid, Meperidine — Administration of meperidine for labor analgesia.
Drug: Labor augmentation, Oxytocin — Oxytocin infusion for augmentation of labor.
  Arms: Spontaneous labor arm
Drug: Labor induction, Oxytocin — Oxytocin infusion for induction of labor.
  Arms: Induced labor arm
Drug: Cervical ripening, labor induction, Dinoprostone — Administration of dinoprostone pessary for cervical ripening and labor induction.
  Arms: Induced labor arm

SUMMARY:
Primary aim of this study is to analyse contemporary labor patterns by measuring rate of dilatation and head descent via transperineal ultrasonography. Labor curves will be generated using data regarding rate of dilatation, head-descent obtained via transperineal ultrasonography. Factors which are known to effect duration of labor will be taken into account.

DETAILED DESCRIPTION:
Intrapartum sonography is rapidly advancing field in the management of obstetrics labor. Traditional approach to labor management consists evaluation of cervical dilatation, head position and head descent via digital examinations. Rate of progress is evaluated using data of available labor curves. Unsatisfactory progression is either treated with labor augmentation or cesarean section depending on the degree and duration of labor retardation. Transperineal ultrasonography is able to assess cervical dilatation, fetal head descent and head position. Data obtained from analysis of labor via transperineal ultrasonography is not available. This research's primary aim is to generate labor curves using data obtained via ultrasonographic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancies
* Spontaneous labor
* Induced labor

Exclusion Criteria:

* Preterm pregnancy
* Previous cesarean section
* Fetal presentation anomalies (breech etc.)
* 5th minute APGAR score lower than 7
* Instrumental delivery (forceps or vacuum use)
* Labor management that is not in accordance with "Safe Prevention of the Primary Cesarean Delivery" guideline by American College of Obstetrics and Gynecology.
* Fetus suffering visible birth trauma (laceration, fracture etc.)

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Duration of active labor | From time of initial admission until the time of birth, up to 36 hours
  Duration of active labor will be calculated in minutes, in a reverse fashion, beginning from time of birth and going back to first time of measurement.
Rate of cervical dilatation advancement as measured by transperineal ultrasonography | From time of initial admission until the time of birth, up to 36 hours
  Rate of cervical dilatation assessment will be measured in millimetres/hour in a reverse fashion beginning from the time when maximum dilatation is achieved and going back to time of first measurement.
Rate of angle of progression advancement as measured by transperineal ultrasonography | From time of initial admission until the time of birth, up to 36 hours
  Rate of angle of progression advancement will be measured in metric degree in a reverse fashion beginning from the last measurement taken and going back to first measurement taken.

SECONDARY OUTCOMES:
Effect of amniotomy on duration of active labor | From time of initial admission until the time of birth, up to 36 hours
  Effect of amniotomy on the duration of labor will be assessed in minutes by analysing the different time points in different labor processes when amniotomy has taken place.

CONTACTS AND LOCATIONS:
Overall Officials: Acar F Koc, Professor, Study Director — Department of Obstetrics and Gynecology, Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Department of Obstetrics and Gynecology, Ankara, Turkey (Türkiye)